CLINICAL TRIAL: NCT01121796
Title: Influence of Vitamin D on Inflammatory Bowel Disease Remission
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Hillel Yaffe Medical Center (Other Government)
Collaborators: Technion, Israel Institute of Technology (Other)
Responsible Party: Dr. Zvi Fireman, Director Gastroenterology Institute, Hillel Yaffe Medical Center
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: HY100510
Record Dates: First submitted 2010-05-10; First posted 2010-05-12 (Estimated); Last update posted 2010-05-12 (Estimated); Status verified 2010-05

CONDITIONS: Inflammatory Bowel Disease
MeSH Terms: conditions — Inflammatory Bowel Diseases | interventions — Vitamin D; Water; Milk

STUDY DESIGN:
Who Masked: Participant, Care Provider

ARMS (3):
- Vitamin D (Active Comparator)
  Interventions: Dietary Supplement: Vitamin D
- Placebo (Placebo Comparator)
  Interventions: Other: Water or milk
- Unique vehicle for Vitamin D supplementation (Active Comparator)
  Interventions: Dietary Supplement: Vitamin D enriched milk

INTERVENTIONS:
Dietary Supplement: Vitamin D
  Arms: Vitamin D
Other: Water or milk
  Arms: Placebo
Dietary Supplement: Vitamin D enriched milk
  Arms: Unique vehicle for Vitamin D supplementation

SUMMARY:
Vitamin D has been shown to influence a multitude of systems. We intend to see whether different types of Vitamin D supplements have an effect on inflammatory bowel disease.

ELIGIBILITY:
Inclusion Criteria:

* Mild to moderate inflammatory bowel disease

Exclusion Criteria:

* Hypersensitivity to milk products

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2010-06; Primary Completion 2011-06 (Estimated)

PRIMARY OUTCOMES:
Inflammatory disease remission | One year

CONTACTS AND LOCATIONS:
Locations (1):
- Hillel Yaffe Medical Center, Hadera, Israel